CLINICAL TRIAL: NCT04811079
Title: The Role of Spectral Filtering in a Spectrally Adjustable Ocular Photosensitivity Analyzer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-6402
Record Dates: First submitted 2021-03-22; First posted 2021-03-23 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Photosensitivity
MeSH Terms: conditions — Photosensitivity Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Spectacle Filter Sequence 1 (Experimental): (419nm, 437nm, 373nm, 456nm, 476nm) Eligible subjects will be enrolled in Spectacle Filter Sequence 1.
  Interventions: Other: 419 nm Spectacle Filter; Other: 437 nm Spectacle Filter; Other: 456 nm Spectacle Filter; Other: 476 nm Spectacle Filter; Other: 373 nm Spectacle Filter
- Spectacle Filter Sequence 2 (Experimental): (437nm, 456nm, 419nm, 476nm, 373nm) Eligible subjects will be enrolled in Spectacle Filter Sequence 2.
  Interventions: Other: 419 nm Spectacle Filter; Other: 437 nm Spectacle Filter; Other: 456 nm Spectacle Filter; Other: 476 nm Spectacle Filter; Other: 373 nm Spectacle Filter
- Spectacle Filter Sequence 3 (Experimental): (456nm, 476nm, 437nm, 373nm, 419nm) Eligible subjects will be enrolled in Spectacle Filter Sequence 3.
  Interventions: Other: 419 nm Spectacle Filter; Other: 437 nm Spectacle Filter; Other: 456 nm Spectacle Filter; Other: 476 nm Spectacle Filter; Other: 373 nm Spectacle Filter
- Spectacle Filter Sequence 4 (Experimental): (476nm, 373nm, 456nm, 419nm, 437nm) Eligible subjects will be enrolled in Spectacle Filter Sequence 4.
  Interventions: Other: 419 nm Spectacle Filter; Other: 437 nm Spectacle Filter; Other: 456 nm Spectacle Filter; Other: 476 nm Spectacle Filter; Other: 373 nm Spectacle Filter
- Spectacle Filter Sequence 5 (Experimental): (373nm, 419nm, 476nm, 437nm, 456nm) Eligible subjects will be enrolled in Spectacle Filter Sequence 5.
  Interventions: Other: 419 nm Spectacle Filter; Other: 437 nm Spectacle Filter; Other: 456 nm Spectacle Filter; Other: 476 nm Spectacle Filter; Other: 373 nm Spectacle Filter
- Spectacle Filter Sequence 6 (Experimental): (476nm, 456nm, 373nm, 437nm, 419nm) Eligible subjects will be enrolled in Spectacle Filter Sequence 6.
  Interventions: Other: 419 nm Spectacle Filter; Other: 437 nm Spectacle Filter; Other: 456 nm Spectacle Filter; Other: 476 nm Spectacle Filter; Other: 373 nm Spectacle Filter
- Spectacle Filter Sequence 7 (Experimental): (373nm, 476nm, 419nm, 456nm, 437nm) Eligible subjects will be enrolled in Spectacle Filter Sequence 7.
  Interventions: Other: 419 nm Spectacle Filter; Other: 437 nm Spectacle Filter; Other: 456 nm Spectacle Filter; Other: 476 nm Spectacle Filter; Other: 373 nm Spectacle Filter
- Spectacle Filter Sequence 8 (Experimental): (419nm, 373nm, 437nm, 476nm, 456nm) Eligible subjects will be enrolled in Spectacle Filter Sequence 8.
  Interventions: Other: 419 nm Spectacle Filter; Other: 437 nm Spectacle Filter; Other: 456 nm Spectacle Filter; Other: 476 nm Spectacle Filter; Other: 373 nm Spectacle Filter
- Spectacle Filter Sequence 9 (Experimental): (437nm, 419nm, 456nm, 373nm, 476nm) Eligible subjects will be enrolled in Spectacle Filter Sequence 9.
  Interventions: Other: 419 nm Spectacle Filter; Other: 437 nm Spectacle Filter; Other: 456 nm Spectacle Filter; Other: 476 nm Spectacle Filter; Other: 373 nm Spectacle Filter
- Spectacle Filter Sequence 10 (Experimental): (456nm, 437nm, 476nm, 419nm, 373nm) Eligible subjects will be enrolled in Spectacle Filter Sequence 10.
  Interventions: Other: 419 nm Spectacle Filter; Other: 437 nm Spectacle Filter; Other: 456 nm Spectacle Filter; Other: 476 nm Spectacle Filter; Other: 373 nm Spectacle Filter

INTERVENTIONS:
Other: 419 nm Spectacle Filter — TEST
Other: 437 nm Spectacle Filter — TEST
Other: 456 nm Spectacle Filter — TEST
Other: 476 nm Spectacle Filter — TEST
Other: 373 nm Spectacle Filter — CONTROL

SUMMARY:
This is a 6-visit, single-center, non-dispensing, randomized, single-masked, 5×5 crossover study. Subjects will participate in 6 scheduled over the duration of approximately 10.5 months.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all of the following criteria to be enrolled in the study:

  1. The subject must read and sign the Informed Consent form.
  2. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
  3. Healthy adult males or females age ≥18 and ≤30 years of age.
  4. Normal color vision as measured using the Ishihara 38-plate test.
  5. Normal stereopsis as measured by a suitable test.
  6. Auto-refraction must show a spherical component of -2.00 through +2.00 D, and a cylindrical component of 0.00 through 1.50 D.
  7. The subject's distance refractive sphere must be between -2.00 and +2.00 D in each eye.
  8. The subject's distance refractive cylinder must be ≤ 1.50 D in each eye.
  9. The subject must have unaided distance Snellen visual acuity of 20/200 or better for each eye.
  10. The subject must have best corrected distance Snellen visual acuity of 20/25 or better for each eye.

      Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Currently pregnant or lactating (subjects who become pregnant during the study will be discontinued).
  2. History of refractive surgery or other ocular surgery.
  3. Employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
  4. Subjects that participated in the pilot study CR-6318.
  5. Systemic conditions or the use of medications that the investigator believes will contraindicate participation in this study.
  6. Abnormal Level 3 neuro-ophthalmology exam including crystalline lens clarity Grade 3 or worse (Lens Opacities Classification System).
  7. Any Grade 3 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA Slit Lamp Classification Scale.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2021-07-14 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
Visual Photosensitivity Threshold (VPT) | at approximately 2-week follow-up
  VPT will measured via the SAOPA instrument. VPT is the point at which a sensation of pain or discomfort occurs when the intensity of light is gradually increased from a low level. Subject's discomfort responses will be indicated via a button press. Testing is complete when 10 response reversals are acquired.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (1):
- University of Miami Health - Bascom Palmer Eye Institute, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu